CLINICAL TRIAL: NCT03481049
Title: Novel EtG-Based Contingency Management for Alcohol in the Severely Mentally Ill
Brief Title: Individualizing Incentives for Alcohol in the Severely Mentally Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael McDonell, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16326; R01AA022070 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2018-03-29 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder; Alcohol Dependence
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual CM (Experimental): Participants will earn at least 3 prize draws each time they submit an alcohol negative urine samples during weeks 5-20, plus treatment as usual
  Interventions: Behavioral: Usual CM
- High-Magnitude CM (Experimental): Participants will earn twice as many prize draws than those in the Usual CM for alcohol abstinence during weeks 5-20, plus treatment as usual.
  Interventions: Behavioral: High-Magnitude CM
- Shaping CM (Experimental): Participants will earn prize draws for light drinking during weeks 5-8 instead of alcohol abstinence and will then earn prize draws for abstinence during weeks 9-20, plus treatment as usual.
  Interventions: Behavioral: Shaping CM

INTERVENTIONS:
Behavioral: Usual CM — Behavioral reinforcement for alcohol abstinence
  Arms: Usual CM
Behavioral: High-Magnitude CM — Behavioral reinforcement for alcohol abstinence
  Arms: High-Magnitude CM
Behavioral: Shaping CM — Behavioral reinforcement for alcohol abstinence
  Arms: Shaping CM

SUMMARY:
The investigators will evaluate the efficacy of a 2 various contingency management (CM) interventions (High-Magnitude CM, Shaping CM) for treating heavy drinking among individuals with serious mental illness and alcohol dependence who are seen within the context of a community mental health center setting. Participants will be 400 adults diagnosed with serious mental illness and alcohol dependence and those who demonstrate heavy drinking during the first 4 weeks will be randomized to receive treatment conditions.

DETAILED DESCRIPTION:
The objective of this study is to determine whether modifications to a CM intervention improve outcomes and reduce costs in heavy drinkers with serious mental illness using alcohol biomarker ethyl glucuronide (EtG) to test of alcohol abstinence. In CM, patients receive tangible rewards for demonstrating drug abstinence.

The investigators propose to examine whether 2 strategies - 1. Increasing reinforcer magnitude (High-Magnitude CM) or 2. Reinforcing light drinking before reinforcing abstinence (Shaping CM) - can improve outcomes in heavy drinkers with serious mental illness. The investigators will compare the efficacy of these 2 approaches to Usual CM in heavy drinkers with serious mental illness.

A total of 400 participants receiving treatment as usual at 2 treatment agencies will take part in a 4-week induction period. Participants (n=240) who attain a mean EtG > 349 ng/mL (heavy drinking) during the induction period will be randomized to either a) 4 months of standard-magnitude CM for submitting alcohol-abstinent EtG samples (EtG < 150 ng/mL) (Usual CM), b) 4 months of high-magnitude CM for submitting alcohol-abstinent EtG samples (High-Magnitude CM), or c) 1 month of CM for submitting alcohol samples that indicate light drinking (EtG < 500 ng/mL), followed by 3 months of CM for submitting alcohol-abstinent EtG samples (Shaping CM). The primary outcome will be EtG-verified alcohol abstinence during the last 3 months of treatment (when all reinforcement is contingent on abstinence) and during 12 months of follow-up.

The investigators will also examine group differences in secondary outcomes, conduct a comprehensive economic analysis, and determine whether variables that make up the NIAAA Addictions Neuroclinical Assessment (ANA) model moderate alcohol abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years.
2. 4 or more standard drinks for females (AFAB)/ 5 or more standard drinks for males (AMAB) on 5 or more occasions in the past 30 days.
3. DSM-5 diagnosis of moderate to severe alcohol use disorder.
4. DSM-5 diagnosis of schizophrenia or schizoaffective disorder, bipolar I or II, or recurrent major depressive disorder (>1 episode).

Exclusion Criteria:

1. Current DSM-5 diagnosis of a severe substance use disorder for any substances used within the past 30 days
2. A significant risk of medically dangerous alcohol withdrawal (e.g. a history of seizures in the last 12 months, participant or clinician concern that abstinence will induce dangerous alcohol withdrawal).
3. Any medical/psychiatric condition, or severity of that condition, that in the opinion of the PI, would compromise safe study participation.
4. Inability to provide informed consent as measured by the MacCAT-CR. (e.g. dementia)
5. Pregnant or planning to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G McDonell, PhD, Principal Investigator — Washington State University
Locations (2):
- United States (2):
  - Sound Health, Seattle, Washington
  - WSU Research Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonell MG, Parent S, Jett JD, Keshtkar M, Palmer K, Beck R, Tyutyunnyk D, Williams M, Weeks DL, Chaytor NS, McPherson S, Murphy SM, Ries RK, Roll JM. Testing adaptations to contingency management for alcohol use disorders: A randomized controlled trial. J Consult Clin Psychol. 2025 Aug;93(8):540-550. doi: 10.1037/ccp0000960. Epub 2025 Jun 26. PMID 40569730

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual CM: Participants will earn at least 5 prize draws each time they submit an alcohol negative urine samples during weeks 5-20, plus treatment as usual
  Usual CM: Behavioral reinforcement for alcohol abstinence
- High-Magnitude CM: Participants will earn at least 15 prize draws for alcohol abstinence during weeks 5-20, plus treatment as usual.
  High-Magnitude CM: Behavioral reinforcement for alcohol abstinence
- Shaping CM: Participants will earn prize draws (at least 5) for light drinking during weeks 5-8 instead of alcohol abstinence and will then earn prize draws for abstinence during weeks 9-20, plus treatment as usual.
  Shaping CM: Behavioral reinforcement for alcohol abstinence
- Not Randomized: This is the group of participants who enrolled in the study but were not eligible for randomization. (Randomization criteria included an induction phase average uEtG >349 ng/mL and attendance in the last week of induction.)
Period: Overall Study
Arm/Group | Usual CM | High-Magnitude CM | Shaping CM | Not Randomized
Started | 53 | 54 | 51 | 234
Completed | 41 | 35 | 37 | 0
Not Completed | 12 | 19 | 14 | 234

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual CM | High-Magnitude CM | Shaping CM | Total
Number analyzed (Participants) | 53 | 54 | 51 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.5) | 42.6 (11.7) | 39.2 (12.1) | 40.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 28 | 84
  Male | 25 | 26 | 23 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 2 | 6 | 3 | 11
  White | 45 | 42 | 41 | 128
  More than one race | 2 | 3 | 3 | 8
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use Assessed by Ethyl Glucuronide (EtG) Detection in Urine
Description: Proportion of uEtG negative samples during weeks 5-16 of treatment. (EtG <150 ng/mL = EtG-negative)
Time Frame: During weeks 5 -16 of treatment
Measure: Mean (Standard Deviation); unit: proportion uEtG negative
Groups:
- High-Magnitude CM: Participants will earn at least 15 prize draws than those in the Usual CM for alcohol abstinence during weeks 5-20, plus treatment as usual.
  High-Magnitude CM: Behavioral reinforcement for alcohol abstinence
- Shaping CM: Participants will earn at least 5 prize draws for light drinking during weeks 5-8 instead of alcohol abstinence and will then earn prize draws for abstinence during weeks 9-20, plus treatment as usual.
  Shaping CM: Behavioral reinforcement for alcohol abstinence.
Arm/Group | Usual CM | High-Magnitude CM | Shaping CM
Number analyzed (Participants) | 53 | 54 | 51
proportion uEtG negative | 0.66 (0.25) | 0.65 (0.26) | 0.61 (0.28)

2. Secondary Outcome: Positive and Negative Syndrome Scale
Description: Psychiatric symptomology
Time Frame: At baseline, week 4, 8, 12, 16 through study completion
Reporting Status: Not Posted

3. Secondary Outcome: Urinanalysis for Drug Use
Description: Urine tests for drug use
Time Frame: Baseline, during 4-week induction period and 16 weeks of treatment (repeated measure)
Reporting Status: Not Posted

4. Secondary Outcome: Addiction Severity Index (ASI)
Description: Alcohol and drug addiction severity
Time Frame: Baseline, week 4, 8, 12, 16 through study completion
Reporting Status: Not Posted

5. Secondary Outcome: Alcohol and Cigarette Timeline Followback
Description: Alcohol and Cigarette Use
Time Frame: Baseline, during 4-week induction period and 16 weeks of treatment (repeated measure)
Reporting Status: Not Posted

6. Secondary Outcome: Fagerstrom Test of Nicotine Dependence
Description: Presence and severity of nicotine dependence
Time Frame: Baseline, week 4, 8, 12, 16 through study completion
Reporting Status: Not Posted

7. Secondary Outcome: Housing Timeline FollowBack
Description: Assess homelessness
Time Frame: Baseline, during 4-week induction period, 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

8. Secondary Outcome: Brief HIV Risk Behavior Scale
Description: HIV risk behavior; with a "drug use" subscale measuring 0 - 30 (with lower scores representing better health outcomes related to drug use and higher scores representing poorer health outcomes related to drug use) and a "sexual behavior" subscale measuring 0 - 25 (with lower scores representing better health outcomes related to sexual behavior and higher scores representing poorer health outcomes related to sexual behavior). Both are summed to create a total score ranging from 0 - 55 (with lower totals representing better health outcomes related to HIV risk and higher totals representing poorer health outcomes related to HIV risk)
Time Frame: Baseline, during 4-week induction period, 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

9. Secondary Outcome: NIH Toolbox Emotion Battery
Description: Negative emotionality
Time Frame: Baseline, during 4-week induction period and 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

10. Secondary Outcome: NIH Toolbox Cognition Battery
Description: Executive functioning
Time Frame: Baseline, weeks 20, 47, 71
Reporting Status: Not Posted

11. Secondary Outcome: Obsessive-Compulsive Drinking Scale
Description: Self-report measure of frequency and consequences alcohol-related thoughts and behaviors; Obsessive subscale ranges from 0 - 20 (with lower score representing better health outcomes and higher scores representing poorer health outcomes) Compulsive subscale ranges from 0 -20 (with lower scores representing better health outcomes and higher scores representing poorer health outcomes). Total score (Obsessive + Compulsive sub scales ) ranging from 0 - 40 (with lower totals representing better health outcomes and higher totals representing poorer health outcomes).
Time Frame: Baseline, 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

12. Secondary Outcome: Stimulus-Response Compatibility Task
Description: Cognitive measure of approach-avoidance of alcohol-related cues
Time Frame: Baseline, weeks 20, 47, 71
Reporting Status: Not Posted

13. Secondary Outcome: Stages of Change Readiness and Treatment Eagerness Scale
Description: Motivation to change alcohol use; total scores range from 19 - 95 (with lower totals representing lesser readiness/eagerness for change and higher totals representing greater readiness/eagerness to change)
Time Frame: Baseline, during 4-week induction period and 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

14. Secondary Outcome: Treatment Experiences and Expediencies Questionnaire
Description: Assess drinking goals
Time Frame: Baseline, during 4-week induction period and 16 weeks of treatment (repeated measure) through study completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from the date the participant enrolled in the study (i.e. baseline), through the 1 month induction phase, the 4 month treatment phase, and the 1 year follow-up phase. Therefore, adverse event data was collected for 17 months for each study participant.
Description: The data safety monitoring plan included the standard definitions accepted by clinicaltrials.gov, with the following differences:
  Because inpatient psychiatric or substance abuse treatment can be considered a worsening of a pre-existing condition with this study populations, these events were reported as Adverse Events, not Serious Adverse Events.
  AEs/SAEs were assessed through regularly scheduled questionnaires and assessments.
Groups:
- Shaping CM: Participants will earn prize draws (at least 5) for light drinking during weeks 5-8 and will then earn prize draws for abstinence during weeks 9-20, plus treatment as usual.
  Shaping CM: Behavioral reinforcement for alcohol abstinence
- Not Randomized: Participants who enrolled in the study but were not eligible for randomization. (Eligibility for randomization included an average induction uEtG >349 ng/mL and attendance in last week of induction.)
Arm/Group | Usual CM | High-Magnitude CM | Shaping CM | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54 | 0/51 | 0/234
Serious Adverse Events (participants affected / at risk) | 4/57 | 3/55 | 7/54 | 2/234
Other Adverse Events (participants affected / at risk) | 30/57 | 21/55 | 23/54 | 63/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual CM (N=57) | High-Magnitude CM (N=55) | Shaping CM (N=54) | Not Randomized (N=234)
Inpatient Medical Treatment (General disorders) | 3 (3) | 2 (3) | 6 (7) | 2 (2)
Suicide Attempt Resulting In Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alcohol Withdrawals that lead to hospitalization (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual CM (N=57) | High-Magnitude CM (N=55) | Shaping CM (N=54) | Not Randomized (N=234)
Alcohol related ER Visit (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
ER Visit (General disorders) | 16 (29) | 9 (14) | 12 (17) | 21 (21)
Inpatient Psychiatric Treatment (Psychiatric disorders) | 7 (11) | 1 (1) | 5 (5) | 3 (3)
Inpatient Substance Abuse Treatment (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Jail (Social circumstances) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
SHOT Score >/= 3 (Nervous system disorders) | 2 (4) | 3 (3) | 0 (0) | 5 (6)
Suicide attempt (not hospitalization) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 19 (28) | 12 (17) | 10 (21) | 32 (35)
Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Injuries that were significant, but did not results in visit to emergency department

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03481049/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03481049/ICF_001.pdf